CLINICAL TRIAL: NCT04914182
Title: Effectiveness of Low Power Laser in the Cicatricial Process and Pain Relief in Primiparous People With Spontaneous Perineal Laceration After Normal Delivery
Brief Title: Low Power Laser for Spontaneous Perineal Laceration
Acronym: LASER
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the Pandemic, the recruitment was very slow. We stopped the study and will continue as soon as the Recruiting Centre reopens the LDR.
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Coordinator of the Obstetrical ICU, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LASER
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Perineal Tear
Keywords: perineal; laser; pain; Visual Analog Scale
MeSH Terms: conditions — Pain | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted, participants will be assigned to the intervention group or the control group in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Control sham: To the patients in the control group a sham control will be applied, corresponding to the device only connected, emitting the signal of being "turned on" but without therapeutic effect. The irradiation time and the number of application points will be the same as for the intervention group. The patient will remain masked, and the investigators that will perform the statistical analysis will be masked until the end of the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LASER (Experimental): In the intervention group, the laser will be applied to the points of the edges of the lesion, with a distance of one centimeter between them. The laser will be applied in a punctual way, in points on the edges of the lesion site, with a distance of one centimeter between them. This application will take place three times: six hours after delivery, 24 and 48 hours after delivery.
  Interventions: Radiation: LASER
- CONTROL (Sham Comparator): In the control group, the sham laser will be applied the exact same way as the real laser, to the points of the edges of the lesion, with a distance of one centimeter between them. The sham laser will be applied in a punctual way, in points on the edges of the lesion site, with a distance of one centimeter between them. This application will take place three times: six hours after delivery, 24 and 48 hours after delivery.
  Interventions: Radiation: CONTROL

INTERVENTIONS:
Radiation: LASER — Laser will be applied in specific points for perineal lacerations.
  Arms: LASER
Radiation: CONTROL — A control group of sham laser will create for the patients the impression that laser is being played, with the lights of the instrument of "on mode" turned on, without biological effects.
  Arms: CONTROL

SUMMARY:
Scenario: spontaneous perineal laceration is an injury to the tissue in the perineum region, which can occur during vaginal delivery. The lesion can be classified into four degrees, according to the structures affected, with degrees one and two being more common. Some consequences may arise due to lacerations, such as perineal pain, genito-pelvic pain, in addition to infection, and dehiscence of the lesion, which may last up to one year after delivery. A laser is a form of non-ionizing radiation and when used in the repair process it is capable of generating analgesic, anti-inflammatory, and healing effects. Low-level laser treatment has been used in several areas, promoting cellular and vascular responses capable of accelerating the repair of injured tissue, in addition to pain relief and consequently capable of improving patients' quality of life. Objective: To determine the effects of low-power laser on the acceleration of the healing process and pain relief in primiparous women who had a spontaneous perineal tear, grade one and two, during normal delivery. Methods: a pilot randomized clinical trial will be carried out. Two groups will be divided randomly, one group will receive the application of the laser, and the second group the laser "sham". Data collection will be carried out at the LAbor and delivery rooms of the Instituto de Medicina Integral Prof. Fernando Figueira (IMIP). Primiparous women who had a spontaneous perineal tear, grades one and two, over 18 years of age or younger who are in charge, with a full-term pregnancy, single fetus, cephalic presentation, and who have been admitted to labor at the ANC will be included, excluding patients who are transferred to another sector, those that evolve to a cesarean section or need episiotomy or curettage and, in addition, the presence of infection during childbirth assistance, postpartum hemorrhage and suspected or diagnosed COVID-19. The laser will be applied at three predetermined moments: six hours, 24, and 48 hours after delivery. To evaluate the healing process a REEDA scale and a Peri-rule will be used. The assessment of pain intensity will be through the Visual Analogue Scale (VAS). Ethical Aspects: the research will be submitted to the IMIP Research Ethics Committee and data collection will begin after its approval. All data will be kept confidential and confidential, the participant will be asked to sign the Informed Consent Form before beginning any procedure.

DETAILED DESCRIPTION:
In primiparous women with spontaneous perineal laceration, grade 1 and 2, during normal delivery submitted to the application of low power laser versus "sham" laser:

1. Describe the biological characteristics (age, weight, height, BMI), sociodemographic (marital status, race, years studied, family income, social occupational);
2. Describe the characteristics related to life habits (smoking, activity physical, pelvic physiotherapy during pregnancy, Pilates during pregnancy, yoga during pregnancy);
3. Describe the previous gynecological and obstetric characteristics (number of pregnancies, type of previous births, number of abortions, suture in childbirth current) and obstetric (prenatal consultations, number of prenatal consultations, gestational age, gestational weight gain, use of oxytocin, use of analgesia, blood flow guidance, position during the second period of childbirth, hours labor, instrumental delivery, birth weight, head circumference of the newborn, shoulder dystocia, perineal laceration, the severity of lacerations, laceration extension, postpartum perineal pain);
4. Compare the parameters of REEDA, such as redness, edema, bruising, secretion and approximation of the edges at each intervention and in the range of seven and 42 days after laser application;
5. Compare the frequency of perineal pain and genito-pelvic pain at each intervention and between seven and 42 days after laser application;
6. Compare the measurement of the extent of perineal laceration, using Peri-Rule, the each intervention and in the interval of seven and 42 days after the application of the laser.

Initially, the study will be carried out with 30 women (pilot study) for later the sample calculation will be carried out. A pilot study will be carried out, as, during the search in the database, no studies were found that address the use of low-level laser in spontaneous perineal lacerations, so that sample calculation was carried out.

Randomization for the intervention and control groups will be performed according to a list of random numbers drawn up for that purpose by an employee who does not was involved with data collection, to ensure confidentiality in the allocation. From this list, sealed and opaque envelopes will be prepared, numbered sequentially, with each number, according to the randomization table, corresponds to the patient's allocation to the intervention or control group.

For statistical analysis of the data, the domain statistical program will be used public Epi-info version 7, or higher versions. Tables will be distributed frequency distribution for categorical variables, calculating the mean and deviation standard of quantitative variables. Then, contingency tables will be used to determine the association of the independent variable (laser application) with the independent variables (REEDA scale, perineal pain, genito-pelvic pain). For determination of the strength of association will be calculated as a measure of the risk (RR) and its 95% confidence interval. All p values will be two-tailed and in all stages of the analysis will be considered a level of significance 5%.

ELIGIBILITY:
Inclusion Criteria:

* Deliveries Assisted at the labor and delivery rooms (low risk)
* Spontaneous perineal laceration (grades 1 and 2)
* Primipara
* Full-term pregnancy (37 to 41 weeks and six days)
* Women over the age of 18 or under who are the presence of a responsible party
* cephalic presentation
* Single fetus
* Admitted in labor

Exclusion Criteria:

* Transfer to another sector;
* Performing an episiotomy;
* Evolution to cesarean section;
* Need for curettage;
* Instrumental delivery (use of forceps and vacuum);
* A patient who had the child referred to another sector;
* Shoulder dystocia;
* Change in skin sensitivity;
* Presence of infection during childbirth care;
* Postpartum hemorrhage;
* Suspected or diagnosed with COVID-19

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
SIZE OF LACERATION 6 hours after delivery | 6 HOURS
  Size in centimeters of the perineal laceration, measured by the PERI-RULE 6 hours after delivery
SIZE OF LACERATION 6 hours after delivery | 24 hours after delivery
  Size in centimeters of the perineal laceration, measured by the PERI-RULE 24 hours after delivery
SIZE OF LACERATION 6 hours after delivery | 48 hours after delivery
  Size in centimeters of the perineal laceration, measured by the PERI-RULE 48 hours after delivery
SIZE OF LACERATION AFTER ONE WEEK | 1 WEEK
  Size in centimeters of the perineal laceration, measured by the PERI-RULE one week after delivery
SIZE OF LACERATION AFTER 42 DAYS | 42 DAYS
  Size in centimeters of the perineal laceration, measured by the PERI-RULE after 42 days of delivery

SECONDARY OUTCOMES:
REDNESS AFTER 5 HOURS | 6 hours after delivery
  Redness evaluated with the REEDA (Redness, Oedema, Ecchymosis, Discharge, Approximation) scale with 6 hours after delivery The REEDA scale is a tool that assesses the inflammatory process and tissue healing in the perineal trauma, through the evaluation of five items of healing: redness (hyperaemia), oedema, ecchymosis, discharge and approximation of the wound edges (coaptation). For each assessed item, a score ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
REDNESS AFTER 24 HOURS | 24 hours after delivery
  Redness evaluated with the REEDA scale with 24 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
REDNESS AFTER 48 HOURS | 48 hours after delivery
  Redness evaluated with the REEDA scale with 48 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
REDNESS AFTER 7 DAYS | 7 days
  Redness evaluated with the REEDA scale with 7 DAYS of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
REDNESS AFTER 42 DAYS | 42 days
  Redness evaluated with the REEDA scale with42 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
EDEMA AFTER 6 HOURS | 6 hours after delivery
  EDEMA evaluated with the REEDA scale with 6 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
EDEMA AFTER 24 HOURS | 24 hours after delivery
  EDEMA evaluated with the REEDA scale with 24 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
EDEMA AFTER 48 HOURS | 48 hours after delivery
  EDEMA evaluated with the REEDA scale with 48 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
EDEMA AFTER 7 DAYS | 7 days
  EDEMA evaluated with the REEDA scale with 7 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
EDEMA AFTER 42 DAYS | 42 days
  EDEMA evaluated with the REEDA scale with 42 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
BRUISING AFTER 6 HOURS | 6 hours after delivery
  BRUISING evaluated with the REEDA scale with 6 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
BRUISING FATER 24 HOURS | 24 hours after delivery
  BRUISING evaluated with the REEDA scale with 24 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
BRUISING AFTER 48 HOURS | 48 hours after delivery
  BRUISING evaluated with the REEDA scale with 48 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
BRUISING AFTER 7 DAYS | 7 days
  BRUISING evaluated with the REEDA scale with 7 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
BRUISING AFTER 42 DAYS | 42 days
  BRUISING evaluated with the REEDA scale with 42 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
PRESENCE OF SECRETION AFTER 6 HOURS | 6 hours after delivery
  PRESENCE OF SECRETION evaluated with the REEDA scale with 6 hours after delivery.
  ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
PRESENCE OF SECRETION AFTER 24 HOURS | 24 hours after delivery
  PRESENCE OF SECRETION evaluated with the REEDA scale with 24 hours after delivery.
  ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
PRESENCE OF SECRETION AFTER 48 HOURS | 48 hours after delivery
  PRESENCE OF SECRETION evaluated with the REEDA scale with 48 hours after delivery.
  ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
PRESENCE OF SECRETION AFTER 7 DAYS | 7 days
  PRESENCE OF SECRETION evaluated with the REEDA scale with 7 days of delivery
PRESENCE OF SECRETION AFTER 42 DAYS | 42 days
  PRESENCE OF SECRETION evaluated with the REEDA scale with 42 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
WOUND CLOSURE AFTER 6 HOURS | 6 hours after delivery
  WOUND CLOSURE evaluated with the REEDA scale 6 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
WOUND CLOSURE AFTER 24 HOURS | 24 hours after delivery
  WOUND CLOSURE evaluated with the REEDA scale 24 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
WOUND CLOSURE AFTER 48 HOURS | 48 hours after delivery
  WOUND CLOSURE evaluated with the REEDA scale 48 hours after delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
WOUND CLOSURE AFTER 7 DAYS | 7 days
  WOUND CLOSURE evaluated with the REEDA scale with 7 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
WOUND CLOSURE AFTER 42 DAYS | 42 days
  WOUND CLOSURE evaluated with the REEDA scale with 42 days of delivery. ranging from 0 to 3 can be assigned by the healthcare provider. A higher score indicates a greater level of tissue trauma.
PERINEAL PAIN AFTER 6 HOURS | 6 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 6 hours of delivery (For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
PERINEAL PAIN AFTER 24 HOURS | 24 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 24 hours of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PERINEAL PAIN AFTER 48 HOURS | 48 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 48 hours of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PERINEAL PAIN AFTER 7 DAYS | 7 days of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 7 days of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PERINEAL PAIN AFTER 42 DAYS | 42 days of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 42 days of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PELVIC PAIN AFTER 6 HOURS | 6 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 6 hours of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PELVIC PAIN AFTER 24 HOURS | 24 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 24 hours of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PELVIC PAIN AFTER 48 HOURS | 48 hours of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 48 hours of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PELVIC PAIN AFTER 7 DAYS | 7 days of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 7 days of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]
PELVIC PAIN AFTER 42 DAYS | 42 days of delivery
  PERINEAL PAIN evaluated with the Pain Visual Analog scale with 42 days of delivery For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]

CONTACTS AND LOCATIONS:
Overall Officials: Melania M Amorim, PhD, Study Director — IMIP
Locations (1):
- Maternidade Professor Barros Lima, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No